CLINICAL TRIAL: NCT02115906
Title: Assessment of Changes in Metabolic Activity in Liver & Skeletal Muscle in Patients Suffering From Acromegaly - a 31P/1H Magnetic Resonance Spectroscopy Pilot Study
Brief Title: Assessment of Changes in Metabolic Activity in Liver & Skeletal Muscle in Patients Suffering From Acromegaly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Krebs, ao. Univ. Prof. Dr. med. univ., Medical University of Vienna
Other Study IDs: THIGHT_2
Record Dates: First submitted 2014-04-11; First posted 2014-04-16 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Acromegalic patients: Acromegalic patients before and after initiation of individual therapy will be investigated by 1H/31P magnetic resonance spectroscopy, thyroid sonography and oral glucose tolerance testing
  Interventions: Other: 1H/31P Magnetic Resonance Spectroscopy; Other: oral glucose tolerance testing; Other: Thyroid sonography
- Healthy control subjects: Age and Body mass index matched control subjects will be investigated by 1H/31P magnetic resonance spectroscopy and oral glucose tolerance testing
  Interventions: Other: 1H/31P Magnetic Resonance Spectroscopy; Other: oral glucose tolerance testing

INTERVENTIONS:
Other: 1H/31P Magnetic Resonance Spectroscopy — The 31P-MRS examinations will be performed in a 7 T MR system (Siemens Healthcare, Erlangen, Germany) using a double-tuned (31P/1H) surface coil (Rapid Biomedical Ltd, Rimpar, Germany), with a diameter of 10 cm. Participants will be investigated lying in lateral position with the right lobe of the liver positioned over the coil.
Other: oral glucose tolerance testing — In patients without overt diabetes, glucose tolerance will be assessed by an oral glucose tolerance test, routinely performed at the outpatients clinic. The test will be performed in the morning after an overnight fast of at least 8 hours. Blood will be drawn via a catheter placed in an antecubital vein of one arm. Blood samples for the assessment of glucose, insulin, C-peptide, free fatty acids and growth hormone will be drawn at baseline as well as 30, 60, 90 and 120 minutes after ingestion of 75g glucose in a solution.
  Concentrations of glucose, insulin and C-peptide will be used to derive parameters of insulin secretion and insulin sensitivity by mathematical modelling.
Other: Thyroid sonography — In acromegalic patients thyroid morphology will be assessed at the outpatient clinic of the Division of Endocrinology and Metabolism, using standard ultrasound technique. Measurements will be performed by a well- experienced physician at baseline and at each follow up examination in an out-patient care setting.
  Groups: Acromegalic patients

SUMMARY:
Growth hormone (GH) plays a pivotal role in the regulation of body composition including ectopic lipid deposition in insulin sensitive organs like liver and skeletal muscle. Recent evidence indicates that the GH-IGF1 axis affects body composition via regulating mitochondrial oxidation capacity.

Thus, excessive GH secretion by a pituitary adenoma (Acromegaly) might be accompanied by increased mitochondrial activity leading to inappropriately low intracellular lipid depots, especially in metabolically active tissue like liver and skeletal muscle.

This study aims to assess metabolic activity and intracellular lipid content in skeletal muscle and liver in patients suffering from acromegaly compared to controls by 31P/1H Magnetic resonance spectroscopy before and in follow up examinations 3, 6 and 12 months after initiation of GH lowering treatments including surgery, somatostatinanalogs or pegvisomant, as well as oral glucose tolerance tests at each examination to assess treatment responses and calculate validated parameters for insulin sensitivity and resistance.

DETAILED DESCRIPTION:
Background: Growth hormone (GH) plays a pivotal role in the regulation of body composition including ectopic lipid deposition in insulin sensitive organs like liver and skeletal muscle. Direct inhibition of growth hormone action by a receptor antagonist has been shown to induce hepatic steatosis and growth hormone replacement decreases liver fat content in obese humans. Of note, recent evidence indicates that the GH-IGF1 axis affects body composition via regulating mitochondrial oxidation capacity.

Hypothesis: Direct and/or indirect effects of GH on mitochondrial function might mediate the changes in body composition and lipid deposition. Thus, excessive GH secretion by a pituitary adenoma (Acromegaly) might be accompanied by increased mitochondrial activity leading to inappropriately low intracellular lipid depots, especially in metabolically active tissue like liver and skeletal muscle.

Aim: Assessment of metabolic activity and intracellular lipid content in skeletal muscle and liver in patients suffering from acromegaly compared to controls.

Methods: Non-interventional study:

* 31P/1H Magnetic resonance spectroscopy before and in follow up examinations 3, 6 and 12 months after initiation of GH lowering treatments including surgery, somatostatinanalogs or pegvisomant.
* oral glucose tolerance tests at each examination to assess treatment responses and calculate validated parameters for insulin sensitivity and resistance.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-75 years

Exclusion Criteria:

* (known) overt diabetes mellitus
* known coronary artery disease (history of myocardial infarction or angina pectoris)
* acute or chronic (inflammatory, metabolic [hyperlipidemia, arterial hypertension, thyroid disorder]) disease (healthy controls)
* intake of medication potentially affecting glucose or lipid metabolism
* metal devices or other magnetic material in or on the subjects body which will be hazardous for NMR investigation [heart pacemaker, brain (aneurysm) clip, nerve stimulators, electrodes, ear implants, post coronary by-pass graft (epicardial pace wires), penile implants, colored contact lenses, patch to deliver medications through the skin, coiled spring intrauterine device, vascular filter for blood clots, orthodontic braces, shunt- spinal or ventricular, any metal implants (rods, joints, plates, pins, screws, nails, or clips without MR-authorization), embolization coil, or any metal fragments or shrapnel in the body].
* tendency toward claustrophobia
* severe liver disorders (plasma transaminases elevated > 3fold)
* any acute inflammatory disease within 2 weeks prior the study
* pregnancy
* nursing
* clinically relevant anemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: acromegalic patients and healthy controls matched for sex, age and body mass index
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Changes in hepatic energy metabolism | before & 3,6,9, and 12 months after initiation of therapy
  The 31P-MRS examinations will be performed in a 7 T MR system (Siemens Healthcare, Erlangen, Germany) using a double-tuned (31P/1H) surface coil (Rapid Biomedical Ltd, Rimpar, Germany), with a diameter of 10 cm.

SECONDARY OUTCOMES:
Changes in hepatic lipid content | before, as well as 3,6,9 &12 months after initiation of therapy
  Hepatic lipid content will be assessed using localized single voxel 1H MRS as published by our study group. STEAM sequence (VOI= 3×3×3 cm3; TE= 30, 50, 70, 120 ms; NA= 4 for each TE) data acquisition will be performed during repetitive single breath holds. Hepatocellular lipid (HCL) content will be calculated from ration of summed area of methylene and methyl resonance to that of water following the individual spin-spin relaxation correction as per cent of total tissue MRS signal (water + methylene + methyl).

OTHER OUTCOMES:
Changes in skeletal muscle energy metabolism | before, as well as 3,6,9 and 12 months after initiation of therapy
  Resting-state ATP turnover will be measured using a ST experiment. The subjects will be lying in a supine position with the surface coil fixed underneath the right calf muscle. Baseline intramyocellular concentrations of phosphorous metabolites will be assessed based on T1 corrected partially relaxed baseline spectra (TR, 15 s; 16 averages). The exchange between γ-ATP and PCr (i.e., CK reaction), and between γ-ATP and Pi (i.e., ATP- synthesis) will be investigated.
Changes in skeletal muscle lipid content | before, as well as 3,6,9 and 12 months after initiation of therapy
  Intramyocellular lipid content will be assessed using localized single voxel 1H MRS as published by our studygroup[34]. STEAM sequence (VOI= 12x12x12 mm3; TE= 20 ms; TR= 4 sec, NA= 16) data acquisition will be performed in two volumes of interest positioned in soleus and tibialis anterior muscle. Separate spectra without water signal suppression (NA= 4) will be obtained from both muscle groups. Intramyocellular lipid content (IMCL) content will be calculated from ratio of area of methylene (1.25 ppm) to that of water following the individual spin-spin relaxation correction as per cent of tissue water MRS signal.
Changes in thyroid morphology | before and 12 months after initiation of individual therapy
  In acromegalic patients thyroid morphology will be assessed at the outpatient clinic of the Division of Endocrinology and Metabolism, using standard ultrasound technique. Measurements will be performed by a well- experienced physician at baseline and at each follow up examination in an out-patient care setting.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Krebs, MD, Prof., Principal Investigator — Medical University of Vienna, Währinger Gürtel 18-20, 1090 Vienna, Austria
Locations (1):
- Medical University Of Vienna, Department of Internal Medicine III, Vienna, Vienna, Austria

REFERENCES:
- [Background] Valkovic L, Gajdosik M, Traussnigg S, Wolf P, Chmelik M, Kienbacher C, Bogner W, Krebs M, Trauner M, Trattnig S, Krssak M. Application of localized (3)(1)P MRS saturation transfer at 7 T for measurement of ATP metabolism in the liver: reproducibility and initial clinical application in patients with non-alcoholic fatty liver disease. Eur Radiol. 2014 Jul;24(7):1602-9. doi: 10.1007/s00330-014-3141-x. Epub 2014 Mar 20. PMID 24647824